CLINICAL TRIAL: NCT04429659
Title: Changes in Refractive Error in Patients With Both Partially Refractive Esotropia and Amblyopia
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Other Study IDs: Sakarya strabismus
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Refractive Errors; Esotropia; Amblyopia Strabismic
MeSH Terms: conditions — Refractive Errors; Esotropia; Amblyopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1, patients with amblyopia and partially refractive ET: children with both amblyopia and partially refractive accommodative esotropia
- Group 2, patients with refractive ET: children with refractive esotropia

SUMMARY:
To investigate changes in refractive errors and evaluate clinical outcomes of strabismus surgery in patients with both amblyopia and partially refractive esotropia (PAET).Amblyopic patients with PAET were enrolled. Non-amblyopic patients with full refractive accommodative esotropia (RAET) were included in the study as a control group. Preoperative and postoperative best corrected visual acuity (BCVA), spherical equivalent (SE), astigmatism, stereoacuity and deviations at near and distance were evaluated and statistically compared in the patient group. The mean BCVA, SE, astigmatism were compared between the patient and the control groups.

DETAILED DESCRIPTION:
Purpose: To investigate changes in refractive errors and evaluate clinical outcomes of strabismus surgery in patients with both amblyopia and partially refractive esotropia (PAET).

Material-Method: Amblyopic patients with PAET were enrolled. Non-amblyopic patients with full refractive accommodative esotropia (RAET) were included in the study as a control group. Preoperative and postoperative best corrected visual acuity (BCVA), spherical equivalent (SE), astigmatism, stereoacuity and deviations at near and distance were evaluated and statistically compared in the patient group. The mean BCVA, SE, astigmatism were compared between the patient and the control groups.

ELIGIBILITY:
Inclusion Criteria:

amblyopic children with partially refractive accommodative esotropia as study group non- amblyopic children with fully refractive accommodative esotropia as control group

-

Exclusion Criteria:

Systemic diseases Neurological disorders and diseases Additional ocular diseases

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: study population was composed of amblyopic children with partially refractive ET.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
spherical equivalent | 36 months
  spherical error plus half of the cylindirical error measured by retinoscopy, diopter
cylindirical error | 36 months
  cylindirical error measured by retinoscopy, diopter

CONTACTS AND LOCATIONS:
Overall Officials: Burcin Cakir, MD, Study Chair — Sakarya University
Locations (1):
- Sakarya University Ophthalmology Department, Sakarya, Turkey (Türkiye)